CLINICAL TRIAL: NCT00004328
Title: Phase II Study of the Pathophysiology and Treatment With Enalapril and Polystyrene Sulfonate for Pseudohypoaldosteronism, Type I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11883; UTMB-403
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Pseudohypoaldosteronism
Keywords: endocrine disorders; pseudohypoaldosteronism; rare disease
MeSH Terms: conditions — Pseudohypoaldosteronism; Endocrine System Diseases; Rare Diseases | interventions — Enalapril; polystyrene sulfonic acid

INTERVENTIONS:
Drug: enalapril
Drug: polystyrene sulfonate

SUMMARY:
OBJECTIVES: I. Establish the sodium and potassium intake that will maintain a normovolemic state in a patient with pseudohypoaldosteronism.

II. Determine the effect of extracellular fluid volume and serum potassium manipulations on exercise tolerance, cardiac function, and endurance.

III. Investigate pharmacologic methods of limiting excretion of sodium in urine and sweat.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Sodium and potassium intake resulting in normalization of serum electrolytes and markers of extracellular volume are determined at baseline. A trial diet is then prescribed, with adjustments made to achieve a steady state with normal serum electrolytes. Exercise tolerance and muscle function are evaluated at steady state.

Sodium and potassium are sequentially manipulated with diet, enalapril, and polystyrene sulfonate. Exercise tolerance is evaluated during each diet period.

A treatment plan to maintain electrolyte balance is developed. The patient is followed monthly for 3 to 6 months, then every 3 months for up to 3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Pseudohypoaldosteronism

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1
Dates: Start 1992-12

CONTACTS AND LOCATIONS:
Overall Officials: Bruce S. Keenan, Study Chair — University of Texas